CLINICAL TRIAL: NCT06799741
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Compare the Safety and Efficacy of 3 Dose Levels of AV-1 in Healthy Adults Challenged With a Controlled Human Infection Strain of DENV-3
Brief Title: A Study to Evaluate the Safety and Efficacy of AV-1 Against Dengue Virus 3 (DENV-3) Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbViro LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV1-PPD-0006
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: DENV-3 Controlled Human Infection Model
Keywords: Healthy Volunteers; Monoclonal antibody; AV-1; Safety; Dengue; Efficacy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1A prophylaxis (Experimental)
  Interventions: Drug: AV-1 100 mg; Drug: Placebo
- Group 2A prophylaxis (Experimental)
  Interventions: Drug: AV-1 300 mg; Drug: Placebo
- Group 3A prophylaxis (Experimental)
  Interventions: Drug: AV-1 900 mg; Drug: Placebo
- Group 1B treatment (Experimental)
  Interventions: Drug: AV-1 100 mg; Drug: Placebo
- Group 2B treatment (Experimental)
  Interventions: Drug: AV-1 300 mg; Drug: Placebo
- Group 3B treatment (Experimental)
  Interventions: Drug: AV-1 900 mg; Drug: Placebo

INTERVENTIONS:
Drug: AV-1 100 mg — human monoclonal antibody (mAb) intravenous solution
  or
  Arms: Group 1A prophylaxis; Group 1B treatment
Drug: AV-1 300 mg — human monoclonal antibody (mAb) intravenous solution
  or
  Arms: Group 2A prophylaxis; Group 2B treatment
Drug: AV-1 900 mg — human monoclonal antibody (mAb) intravenous solution
  or
  Arms: Group 3A prophylaxis; Group 3B treatment
Drug: Placebo — (0.9% saline intravenous solution) 12:2

SUMMARY:
The goal of this clinical trial is to determine the prophylactic and therapeutic effect of AV-1 in healthy adults using a DENV-3 controlled human infection model (CHIM)

ELIGIBILITY:
Inclusion Criteria:

* Males or nonpregnant, nonlactating females who were assigned males and females at birth, of any race, between 18 and 55 years of age
* Body mass index between 18.5 and 34.9 kg/m², inclusive, at Screening or Study Day -1 (Cohort A) or Study Day 0 (Cohort B)
* Normal 12-lead electrocardiogram (ECG). Normal ECG is defined as the absence of:

  1. QTcF >450 ms in men or >460 ms in women
  2. PR >220 ms ventricular or atrial premature contractions in couplets or higher in grouping
  3. Complete left or right bundle branch block
  4. 2nd or 3rd degree atrioventricular block
  5. Sustained ventricular or atrial arrhythmia
  6. ST elevation consistent with cardiac ischemia
  7. Potential subjects with non-clinical sinus arrhythmia could be included in the study
* Subjects in good health as determined by past medical history, medication use, physical examination, vital signs, and 12-lead ECG at Screening
* Females of childbearing potential must agree to use effective contraception through study duration

  1. Reliable methods of contraception include: long acting, reversible contraception (LARC), hormonal birth control* (implantable device, hormonal patch, hormonal vaginal ring, oral contraception, Depo-Provera injection, etc.), surgical sterilization (hysterectomy, tubal ligation, or tubal coil at least 90 days prior to Investigational Product [IP] dosing)
  2. Must agree to not donate ova or oocytes during the study
  3. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea without an alternative medical cause for amenorrhea, with follicle-stimulating hormone (FSH) concentration ≥40 mIU/mL at Screening and must have a negative pregnancy test result at Screening and Day-1 (Cohort A) or Day 0 (Cohort B)
  4. Surgically sterile women (defined as those who have had a hysterectomy, bilateral salpingectomy, bilateral oophorectomy, tubal ligation, or an Essure placement with radiological confirmation test at least 90 days after procedure) must have a negative pregnancy test result at Screening and Study Day -1 (Cohort A) or Study Day 0 (Cohort B). *Subjects on hormonal birth control must not be on medications or other agents that decrease the effectiveness of hormonal birth control
* Male subjects having sexual intercourse with biologic females and who are biologically capable of fathering children must agree and commit to use male condoms from Study Day -1 until the follow-up visit on Study Day 155 (± 7). A male subject is considered capable of fathering children even if his sexual partner is sterile or using contraceptives

  a. Male subjects must refrain from sperm donation from Study Day -1 until the follow-up visit on Study Day 155 (± 7)
* Understands study and agrees to and is available for all procedures throughout the study
* Agree to follow study restrictions and are able to sign an informed consent form

Exclusion Criteria:

* Any significant medical condition who, in the opinion of the investigator, would interfere with the ability to participate in the study or increase the risk of participating for that subject based on the Investigator's Brochures and the safety profiles of AV-1 and rDEN3Δ30
* Any psychiatric condition or history of psychiatric condition that, in the opinion of the investigator or sponsor, would interfere with the subject's ability to participate in the study or increase the risk of the participation for that subject
* History of significant alcoholism or drug/chemical abuse within 12 months prior to Study Day -1 that has caused medical, occupational, or family problems as indicated by subject history
* Currently being treated for peptic ulcer disease or Helicobacter pylori or has been treated within the 6 months prior to Day -1
* Confirmed screening laboratory value of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), or serum creatinine. Values of Grade 1 or above for these tests may be repeated once to confirm a Grade 1 or above value. Abnormal laboratory values other than those specified will not be exclusionary if the clinician deems them not clinically significant
* History of or suspected coagulopathy
* Alcohol consumption of >21 units* per week for males and >14 units per week for females (*1 unit of alcohol equals 12 oz [360 mL] beer, 1.5 oz [45 mL] liquor, or 5 oz [150 mL] wine) through Study Day 28
* Positive urine drug screen at Screening for drugs of abuse defined as Amphetamines, Barbiturates, Benzodiazepines, Cocaine Metabolite, Opiates, Oxycodone, Phencyclidine without confirmation of medical need verified by prescription (ie, anxiolytics or pain medications).
* Women with positive pregnancy test at either Screening visit, Study Day -1, or Study Day 0
* Seropositive for Hepatitis B surface antigen (HBsAg) or positive for Hepatitis C RNA at Screening
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including, but not limited to, human immunodeficiency virus infection, or use of anti-cancer chemotherapy or radiation therapy (cytotoxic) in the 3 years prior to Screening
* Plan to travel to an area with active Zika virus (ZIKV) or DENV, transmission during the study or returned from travel to an area with active transmission within 30 days of Screening. (*Refer to the Centers for Disease Control and Prevention [CDC] website for areas with active ZIKV or DENV)
* History of vaccination with a licensed or investigational ZIKV vaccine, DENV vaccine*, yellow fever virus (YFV) vaccine, or Japanese encephalitis vaccine or reportedly diagnosed with a ZIKV or DENV infection or disease. (*Includes subject's verbal history of vaccination or disease).
* Positive serology to DENV, ZIKV, West Nile virus (WNV), YFV, or St. Louis encephalitis virus (SLE) within 60 days of Screening
* History of anaphylaxis to any drug compound, (including citrate or polysorbate), food, or other substance, unless approved by the investigator
* Major non-elective surgery within the last 3 months
* Previously treated with a licensed or investigational monoclonal or polyclonal antibody within the past 18 months prior to Study Day -1
* Received any investigational drug product within that last 28 days of Study Day -1
* Any prohibited medication within the past 28 days or plans to use prohibited medication during the study. Prohibited medications include oral/systemic anti-neoplastic agents, medications/supplements known to alter drug absorption, metabolism, or elimination processes (eg, St. John's wort), immunosuppressive drugs
* Use of any aspirin product in the 7 days prior to Study Day -1 through 14 days post-challenge
* Use of an NSAID from 48 hours prior to challenge through 14 days post-challenge
* Participants who have received or plan to receive any vaccination (live), experimental or otherwise, within the past 28 days or after Study Day -1 and 14 days (2 weeks) for inactivated vaccines and mRNA vaccines
* Has received blood products within 60 days (2 months) prior to Study Day -1 (Cohort A) or Day 0 (Cohort B)
* Has donated or lost in excess of 450 mL of blood or plasma within 56 days (8 weeks) of Study Day -1. The subject must also agree to refrain from donating blood or plasma during the study
* Has poor peripheral venous access during screening
* Has previously completed or was withdrawn from this study
* Is a current study site staff paid entirely or partially by the contract for this study, or staff who are supervised by the principal or sub-investigators
* Subjects, who in the opinion of the investigator, should not participate in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Through day 155 (±7 days)
  Defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related
Severity of AEs | Through day 155 (±7 days)
Incidence of Serious Adverse Events (SAEs) | Through day 155 (±7 days)
  Defined as an AE that is unexpected and serious as determined by the Sponsor
Severity of SAEs | Through day 155 (±7 days)
Anti-AV-1 antibodies (ADA) Immunogenicity Testing | Through day 155 (±7 days)
Frequency of viremia | Through day 155 (±7 days)
  Detected by direct serum titration
Duration of viremia | Through day 155 (±7 days)
  Defined as the time from the first infection to the time of the last infection
Viral load | Through day 155 (±7 days)
  Measured by qRT-PCR
Viral load | Through day 155 (±7 days)
  Measured by plaque assay
Change from baseline values of diastolic blood pressure | Through day 155 (±7 days)
Change from baseline values of systolic blood pressure | Through day 155 (±7 days)
Change in baseline values of temperature | Through day 155 (±7 days)
Change in baseline values of respiration rate | Through day 155 (±7 days)
Change in baseline values of heart rate | Through day 155 (±7 days)

SECONDARY OUTCOMES:
Number of participants with detectable DENV-specific IgM antibodies | Baseline through day 155 (±7 days)
Percentage of participants with detectable DENV-specific IgM antibodies | Baseline through day 155 (±7 days)
Number of participants with detectable anti-DENV NS1 IgG antibodies | Baseline through day 155 (±7 days)
Percentage of participants with detectable anti-DENV NS1 IgG antibodies | Baseline through day 155 (±7 days)
Measure AV-1 concentration in human serum by anti-idiotype enzyme-linked immunosorbent assay (ELISA) | Through day 155 (±7 days)
Area under the serum concentration-time curve (AUC) from time 0 to 48 hours post-dose of AV-1 (AUC0-48) | Up today 155 (±7 days)
AUC from time 0 to infinity of AV-1 (AUC0-inf) | Up to day 155 (±7 days)
AUC from time 0 to the time of the last quantifiable concentration of AV-1 (AUC 0- tlast) | Baseline through day 155 (±7 days)
Maximum observed serum concentration of AV-1 (Cmax) | Baseline through day 155 (±7 days)
Time to Cmax of AV-1 (Tmax) | Baseline through day 155 (±7 days)
Apparent serum terminal elimination half-life of AV-1 (t1/2) | Baseline through day 155 (±7 days)
Total serum clearance of AV-1 (CL) | Baseline through day 155 (±7 days)
Volume of distribution during the terminal phase of AV-1 (Vz) | Baseline through day 155 (±7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Urban Ramstedt, PhD, Study Director — AbViro LLC
Locations (3):
- United States (3):
  - Center for Immunization Research (CIR) JHBSPH, Baltimore, Maryland
  - Center for Immunization Research Inpatient Unit, Baltimore, Maryland
  - UVM Larner College of Medicine Department of MMG, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No